CLINICAL TRIAL: NCT01327443
Title: Exercise Versus Diet in the Treatment of Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamal Ibdah, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1142777
Record Dates: First submitted 2010-11-08; First posted 2011-04-01 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; Weight loss; Exercise; NAS scores; Mitochondrial dysfunction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Weight Loss; Motor Activity; Mitochondrial Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weight loss (Other): 10% weight loss in 24 weeks time period through nutritional counseling.
  Interventions: Behavioral: Weight loss
- Exercise without weight loss (Active Comparator): 24 weeks under direct supervision.
  Interventions: Behavioral: Exercise
- Control (No Intervention): No change in usual exercise levels or food intake.

INTERVENTIONS:
Behavioral: Weight loss — Nutritional counseling
  Arms: Weight loss
Behavioral: Exercise — Under direct supervision
  Arms: Exercise without weight loss

SUMMARY:
The central hypothesis of this proposal is that a reduction in hepatic mitochondrial function is the main pathophysiology behind NAFLD (Non-Alcoholic Fatty Liver Disease) and NASH (Non alcoholic steatohepatitis). The investigators further hypothesize that lifestyle modifications through aerobic exercise training without weight loss or diet-induced weight loss are effective in reducing NAFLD parameters by improving hepatic mitochondrial content and function in human subjects.

The investigators propose a randomized, controlled human clinical trial to compare the effects of aerobic exercise training (without weight loss) versus diet-induced weight loss (without exercise) in individuals who have NAFLD or liver biopsy-confirmed NASH

DETAILED DESCRIPTION:
Fatty Liver Disease) and NASH (Non alcoholic steatohepatitis). The investigators further hypothesize that lifestyle modifications through aerobic exercise training without weight loss or diet-induced weight loss are effective in reducing NAFLD parameters by improving hepatic mitochondrial content and function in human subjects.

The investigators propose a randomized, controlled human clinical trial to compare the effects of aerobic exercise training (without weight loss) versus diet-induced weight loss (without exercise) in individuals who have NAFLD or liver biopsy-confirmed NASH

ELIGIBILITY:
Inclusion Criteria:

* sedentary individual between
* age group 18-60 years old
* elevated Liver Function Tests (LFT's) with fatty liver on ultrasound and biopsy proven NASH

Exclusion Criteria:

* significant history of alcohol consumption > 20 gm/day (> 2 drinks / day)
* evidence of other causes of hepatitis including positive screening B & C, autoimmune hepatitis, hemochromatosis, celiac disease, Wilson's disease, alpha 1 antitrypsin deficiency or medication-induced hepatitis
* Subjects with planned exercise > 30-60 minutes per week
* BMI < 25 or > 44 kg/m2
* clinical or biochemical evidence of decompensated liver disease, advanced cardiac or renal disease
* changes in last 3 months the dose of oral hypoglycemic medication and statin,
* positive stress test
* pregnant women
* demented individuals who cannot give consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
NASH ( Non alcoholic steatohepatitis score) on liver biopsy | baseline and 24 weeks

SECONDARY OUTCOMES:
Liver Function Tests | Baseline and 24 weeks
  ALT/AST.
DXA Scan | Baseline and 24 weeks
Ultrasonographical changes in liver echotexture | Baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Ibdah, MD; PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No